CLINICAL TRIAL: NCT01040026
Title: A Phase I/II Single Center Study to Assess Tolerability and Feasibility of Infusions of Allogeneic Expanded Haploidentical Natural Killer (NK) Cells in Patients Treated With High Dose Melphalan Chemotherapy and Autologous Stem Cell Transplantation for a Multiple Myeloma
Brief Title: Expanded Natural Killer (NK) Cells for Multiple Myeloma Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK_MM_01
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NK cell infusions (Experimental): 10 NK cell infusions day 3-30; Treatment with in vitro expanded haploidentical NK cells
  Interventions: Other: Treatment with in vitro expanded haploidentical NK cells

INTERVENTIONS:
Other: Treatment with in vitro expanded haploidentical NK cells — 10 expanded NK-DLI will be applied at fixed intervals and to each patient within 30 days (3 applications per week, Mo/We/Fr) starting with increasing CD56+CD3- NK cell doses at 3 dose levels (1.5x10e6/kg, 1.5x10e7/kg and 1x10e8/kg) and, if safe, continuing with maximally 7 doses of 1x10e8/kg. Maximal cumulative T-cell dose is fixed at <1x10e5/kg

SUMMARY:
High-dose chemotherapy with melphalan and autologous hematopoietic stem cell transplantation (HSCT) is considered standard treatment for patients with multiple myeloma. While autologous HSCT may induce remission in patients resistant to standard chemotherapy, and has been shown to lead to long-lasting disease control in a subgroup of patients, the procedure is not curative. Given enough time and in the absence of a competing cause of death, all patients eventually relapse after auto-HSCT.

The only potentially curative approach currently available in the treatment of multiple myeloma (MM) is stem cell trans-plantation from an allogeneic donor. Allogeneic HSCT eradicates residual myeloma cells through T-cell mediated graft-versus-tumor effects. Allogeneic HSCT is, however, associated with significant risk of graft-versus-host disease and its use is therefore limited to younger patients with high risk dis-ease. Malignant plasma cells in multiple myeloma are also sensitive to natural killer cell lysis. Natural killer cells do not cause graft-versus-host disease, which has led to interest in their therapeutic use in patients with multiple myeloma.

We have previously shown that immunomagnetic separation of a highly pure NK cell product from a leukapheresis is possible and that these cells can be expanded up to 100-fold in a GMP-compatible setting. The current study aims to test the tolerability and feasibility of infusions of in vitro expanded haploidentical NK cells for patients after melphalan 200mg/m2 high dose chemotherapy and autologous HSCT in 10 patients. If feasible, the data will provide a basis for further prospective studies.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years, with multiple myeloma and indication for an autologous HSCT
* Available related haploidentical donor
* Written informed consent

Exclusion Criteria:

* Patients scheduled for autologous/allogeneic tandem HSCT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Safety of expanded NK cell infusion | One year after infusion.

SECONDARY OUTCOMES:
Treatment efficacy | One year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Passweg, MD, Prof., Principal Investigator — Dep. of Hematology, Petersgraben 4, CH-4031 Basel
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Tschan-Plessl A, Kalberer CP, Wieboldt R, Stern M, Siegler U, Wodnar-Filipowicz A, Gerull S, Halter J, Heim D, Tichelli A, Tsakiris DA, Malmberg KJ, Passweg JR, Bottos A. Cellular immunotherapy with multiple infusions of in vitro-expanded haploidentical natural killer cells after autologous transplantation for patients with plasma cell myeloma. Cytotherapy. 2021 Apr;23(4):329-338. doi: 10.1016/j.jcyt.2020.09.009. Epub 2020 Nov 29. PMID 33268029
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/33268029/